CLINICAL TRIAL: NCT05544799
Title: Case Studies of Patients Who Had Experienced Near Death Experience
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Dong-Yeop Shin, Professor, Seoul National University Hospital
Other Study IDs: K-NDE
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Near Death Experience
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Saliva for DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervension

SUMMARY:
An prospective observational study to interview patients who had near death experiences among those who had received intensive care unit intervention during admission in hematology ward.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥19yrs) who are in admission in the Hematology ward of Seoul National University Hospital, and one of the following conditions.

  1. recovered after cardiopulomary resuscitation
  2. recovered after mechanical ventilator
  3. recovered after ICU care
  4. recovered after emergent operation
  5. recovered after Shock, coma, altered mentality
  6. Other medical conditions approaching death

Exclusion Criteria:

1. Those who do not agree to participate this study
2. Those who can not be interviewed due to insufficient recovery from critical medical problems

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hematologic cancers who are in admission.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of near death experience (NDE) | 5 years
  Incidence of case with NDE scale ≥7 point

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Yeop Shin, MD, PhD, Principal Investigator — Department of Internal Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No